CLINICAL TRIAL: NCT06601647
Title: A Prospective, Randomized, Double-blind Study: Effects of Different Adjuvants Combined With Ropivacaine in Interscalene Block on Postoperative Outcomes After Arthroscopic Rotator Cuff Repair
Brief Title: Efficacy of Different Adjuvants With Ropivacaine in Brachial Plexus Block on Anthroscopic Rotator Cuff Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Hsin-Yi Wang, Doctor, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-07-006C
Record Dates: First submitted 2024-08-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ropivacaine (Active Comparator): 0.6% ropivacaine, control
  Interventions: Procedure: adjuvant type
- ropivacaine + dexamethasone (Experimental): 0.6% ropivacaine + 2mg dexamethasone
  Interventions: Procedure: adjuvant type
- ropivacaine + dexmedetomidine (Experimental): 0.6% ropivacaine + 025ug/kg dexmedetomidine
  Interventions: Procedure: adjuvant type
- ropivacaine + dexamethasone + dexmedetomidine (Experimental): 0.6% ropivacaine + 2mg dexamethasone + 0.25/ug/kg dexmedetomidine
  Interventions: Procedure: adjuvant type

INTERVENTIONS:
Procedure: adjuvant type — ropivacaine combined with adjuvant

SUMMARY:
The pain after shoulder rotator cuff repair surgery is severe due to the inflammatory reaction of tendon repair. Severe pain will reduce the patient's shoulder range of motion and delay functional recovery. The use of powerful analgesics for pain relief may also increase the chance of opiate analgesic-related side effects. Brachial plexus block with local anesthetic is widely used for pain control at the acute stage after shoulder arthroscopic surgery, but the maintenance time is often limited. Ropivacaine is a local anesthetic commonly used for brachial plexus block, and its half-life time is 11.8 hours. Clinical studies showed that using ropivacaine plus adjuvants such as dexamethasone or dexmedetomidine for brachial plexus block significantly extended the block duration, reduced postoperative pain, and reduced the use of opiate analgesics. However, the safest and most effective combination of local anesthetics remains unresolved.

This trial aims to evaluate and compare the effects of brachial plexus block using dexamethasone and dexmedetomidine combined with ropivacaine on postoperative pain control and functional recovery after arthroscopic rotator cuff repair surgery.

DETAILED DESCRIPTION:
Shoulder joint surgery is an orthopedic surgery recognized to cause severe postoperative pain. The pain after shoulder rotator cuff repair surgery is severer than other shoulder joint surgeries due to the inflammatory reaction of tendon repair. Severe pain will reduce the patient's shoulder range of motion and delay postoperative functional recovery, and the use of powerful analgesics for pain relief may also increase the chance of side effects related to opiate analgesics. Therefore, postoperative pain control has become an important clinical issue.

Brachial plexus block with local anesthetic is widely used for pain control at the acute stage after shoulder arthroscopic surgery, but the maintenance time is often limited. Ropivacaine is a local anesthetic commonly used for brachial plexus block, and its half-life time is 11.8 hours. Clinical studies showed that using ropivacaine plus adjuvants such as dexamethasone or dexmedetomidine to perform brachial plexus block significantly extended the block duration, reduced postoperative pain, and reduced the use of opiate analgesics. Brachial plexus block with low-dose dexmedetomidine plus ropicavaine significantly prolonged analgesia by 4 hours (14 hours vs. 10 hours) compared to ropicavaine alone, and reduced the dose of opiate analgesias in the first 24 hours after surgery. Compared to ropicavaine only, low-dose dexamethasone plus ropivacaine effectively extended the analgesic duration by 8 hours (19.7 hours vs. 11.8 hours) and reduced the dose of opioid analgesics within 36 hours after surgery (6.5mg versus 2mg). Meanwhile, continuous administration of ropicavaine through a catheter for brachial plexus block can maintain effective analgesia. However, the safest and most effective combination of local anesthetics remains unresolved.

This trial aims to evaluate and compare the effects of brachial plexus block using adjuvants dexamethasone and dexmedetomidine combined with ropivacaine on postoperative pain control and functional recovery following arthroscopic rotator cuff repair surgery. Specifically, we will examine the effect of dexamethasone or dexmedetomidine alone, and in combination, on the duration of the analgesic effect of ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

* age>=20 years
* scheduled to anthroscopic rotator cuff repair at VGH, Taipei

Exclusion Criteria:

* with central or peripheral neurological disease
* refuse to sign informed consent
* ASA score >=4
* blood oxygen saturation concentration <90% when without using oxygen
* emergent surgery
* unstable vital signs (ie, use of vasopressors or inotropes)
* nasal mucosa damage or a history of nasal or skull base surgery
* not suitable for regional anesthesia (ie, abnormal coagulation function, taking anticoagulants)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-19 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain evaluated by NRS | postoperative 1hr (hour), 6hrs, 12hrs, 18hrs, 24hrs, 36hrs, 48hr; 3days , 7days, 14days, 30days, 60days, 180days
  pain level by Numeric rating scale( 11 points ranging from 0 to 10; higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Yi Wang, MD, PhD, Principal Investigator — VGHTPE
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan